CLINICAL TRIAL: NCT03045835
Title: Baska ® Mask Versus Endotracheal Tube in Laparoscopic Cholecystectomy : A Prospective Randomized Trial
Brief Title: Baska ® Mask Versus Endotracheal Tube in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Ng Ching Choe, MD, MMED (Anaes), University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MREC ID NO: 201713-4728
Record Dates: First submitted 2017-01-25; First posted 2017-02-08 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Laparoscopic Surgery
Keywords: laparoscopic cholecystectomy BASKA mask Endotracheal tube
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BASKA mask (Experimental): Selection of size : size 3 (30-50kg), size 4 (50-70kg), size 5 (70-100kg)
  Interventions: Device: BASKA mask
- Endotracheal intubation (Active Comparator): Selection of size : ID 7.0-7.5mm (women), ID 7.5-8.0mm (men)
  Interventions: Device: Endotracheal intubation

INTERVENTIONS:
Device: BASKA mask — Baska mask will be inserted during induction of anaesthesia and once patient is in an adequate anaesthetic depth
  Arms: BASKA mask
Device: Endotracheal intubation — Endotracheal intubation will be carried out during induction of anaesthesia and once patient is in an adequate anaesthetic depth
  Arms: Endotracheal intubation

SUMMARY:
Baska mask is a new novel supraglottic airway device with many salient features. The investigators aim to determine the benefit of BASKA mask as an effective airway device for laparoscopic surgery, and whether it can even substitute endotracheal intubation, in order to smoothen the surgery and anaesthesia process as well as reduce perioperative complications.

DETAILED DESCRIPTION:
Patient's satisfaction and smooth process is crucial for perioperative care.Conduct of Anaesthesia including choice of airway devices play an important role. Endotracheal intubation has long been regarded as the technique of choice for airway management in laparoscopic surgery. However, there is currently an emerging interest in laryngeal mask as the substitute for endotracheal tube in laparoscopic surgery.

The increased abdominal pressure secondary to gas insufflation in Laparoscopic surgery demands a good supraglottic airway device with features of good seal, aspiration prevention and effective ventilation.

Few studies have evaluated the performance Baska® Mask for various type of surgery and had obtained high "first-attempt" success rate, easy insertion and a good oropharyngeal leak pressure above 30cmH2O with low complications such as sorethroat, dysphonia and dysphagia.

However, study regarding comparison of Baska® mask with endotracheal tube has not been carried out before. Therefore, the investigators would like to evaluate this novel device in comparison with endotracheal tube for laparoscopic surgery in our centre.

This will be a prospective randomized controlled study in University Malaya Medical Centre to compare Baska® mask with the conventional laryngoscope-guided endotracheal intubation for laparoscopic surgeries.

The investigators would like to study the efficacy of this device in term of : time to effective airway insertion, efficacy of airway seal, post-operation device of complications.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years old
* American Society of Anesthesiologists (ASA) physical status I and II BMI ≤ 35
* Laparoscopic cholecystectomy only

Exclusion Criteria:

* Known gastroesophageal reflux
* History of difficult intubation or difficult anaesthesia
* Features of facial, laryngeal and pharyngeal anatomy problem

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Time to effective airway insertion | 1 hour
  defined as time from picking up the airway device (either BASKA mask or Endotracheal tube), insertion and until occurrence of the first square-waveform capnogram

SECONDARY OUTCOMES:
Numbers of attempt of airway device insertion and Ease of insertion | 1 hour
  defined as: 1 - first attempt easy, smooth insertion; 2 - second attempt, insertion with resistance; 3 - three attempts, insertion with difficulty; 4 -failed insertion of the SGAs and need to crossover to ETT group
Gastric distension scoring by surgeon | during operative duration
  on a visual analogue scale 0-10 (Figure 2), where 0 = empty stomach, and 10 = heavy distension that interfered with surgical exposure at a) entry of the laparoscope following peritoneal insufflation and b) immediately before removal of the laparoscope at the end of the surgical procedure
Post operation incidence of complications | from the induction of anaesthesia, until at the postanaesthetic care unit (PACU), assessed up to 24 hours
  patients are assessed for the incidence of sore throat, airway trauma (lip, tongue, teeth, blood-staining on device), nausea, vomiting, airway spasm, aspiration, emergence cough
Hemodynamic changes | after induction of anaesthesia at 1, 2, 3,4,5,10,20,30 minutes; then post extubation at 1 ,2,3,4,5 minutes
  Blood pressure and Heart rate

OTHER OUTCOMES:
oropharyngeal leak pressure (OPL) of the device during operation | during operative duration
  the above pressure is measured by performing the maneuver: the expiratory valve of the anaesthetic machine is closed and with a fixed gas flow of 3 L/min, the airway pressure at which equilibrium is reached is recorded. Maximal allowable airway pressure is 40 cm H2O [ OLP is measured at following timeframe - T1: immediately post intubation; T2 : before CO2 insufflation; T3 : after CO2 insufflation; T4 and beyond : each change of position as required during operation (eg. Trendelenburg, reverse Trendelenburg, left tilt)
peak airway pressure of the device during operation | during operative duration
  the above pressure is recorded from the anaesthetic machine at following timeframe - T1: immediately post intubation; T2 : before CO2 insufflation; T3 : after CO2 insufflation; T4 and beyond : each change of position as required during operation (eg. Trendelenburg, reverse Trendelenburg, left tilt)

CONTACTS AND LOCATIONS:
Overall Officials: CHING CHOE NG, MMED(ANAES), Principal Investigator — UNIVERSITY OF MALAYA MEDICAL CENTRE
Locations (1):
- University Malaya Medical Centre, Petaling Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ng CC, Sybil Shah MHB, Chaw SH, Mansor MB, Tan WK, Koong JK, Wang CY. Baska mask versus endotracheal tube in laparoscopic cholecystectomy surgery: a prospective randomized trial. Expert Rev Med Devices. 2021 Feb;18(2):203-210. doi: 10.1080/17434440.2021.1865796. Epub 2020 Dec 31. PMID 33322949